CLINICAL TRIAL: NCT03609775
Title: A Double-blind, Randomized, Placebo-controlled, Double-dummy, Four-way Crossover Study to Investigate the Drug-drug Interactions Between ACT-541468 and Ethanol in Healthy Subjects
Brief Title: A Study to Investigate the Drug-drug Interactions Between ACT-541468 and Ethanol in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Idorsia Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: ID-078-111
Record Dates: First submitted 2018-07-25; First posted 2018-08-01 (Actual); Last update posted 2018-10-15 (Actual); Status verified 2018-10

CONDITIONS: Healthy
MeSH Terms: interventions — daridorexant; ethanol lumiflavine

STUDY DESIGN:
Intervention Model Description: Double-dummy, four-way crossover study design
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Treatment A (ethanol + ACT-541468) (Experimental): 5 h i.v. ethanol clamp at a level of 0.6 g/L in combination with a single oral dose of ACT-541468 (50 mg)
  Interventions: Drug: ACT-541468; Other: Ethanol 10%
- Treatment B (ethanol placebo + ACT-541468) (Experimental): 5 h i.v. placebo clamp in combination with a single oral dose of ACT-541468 (50 mg)
  Interventions: Drug: ACT-541468; Other: Ethanol placebo
- Treatment C (ethanol + ACT-541468 placebo) (Experimental): 5 h i.v. ethanol clamp at a level of 0.6 g/L in combination with a single oral dose of matching ACT-541468 placebo
  Interventions: Other: ACT-541468 placebo; Other: Ethanol 10%
- Treatment D (ethanol placebo + ACT-541468 placebo) (Experimental): 5 h i.v. placebo clamp in combination with a single oral dose of matching ACT-541468 placebo
  Interventions: Other: ACT-541468 placebo; Other: Ethanol placebo

INTERVENTIONS:
Drug: ACT-541468 — One tablet of 50 mg ACT-541468 will be administered orally.
  Arms: Treatment A (ethanol + ACT-541468); Treatment B (ethanol placebo + ACT-541468)
Other: ACT-541468 placebo — Matching ACT-541468 placebo will be administered orally as 1 tablet.
  Arms: Treatment C (ethanol + ACT-541468 placebo); Treatment D (ethanol placebo + ACT-541468 placebo)
Other: Ethanol 10% — Ethanol 10% w/v solution in 5% glucose will be administered i.v. for 5 h and clamped at an ethanol level of 0.6 g/L.
  Arms: Treatment A (ethanol + ACT-541468); Treatment C (ethanol + ACT-541468 placebo)
Other: Ethanol placebo — Matching placebo for the ethanol infusion (i.e., 5% glucose solution) will be administered i.v. for 5 h.
  Arms: Treatment B (ethanol placebo + ACT-541468); Treatment D (ethanol placebo + ACT-541468 placebo)

SUMMARY:
A study to investigate the drug-drug interactions between ACT-541468 and ethanol in healthy subjects

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent prior to any study-mandated procedure.
* Healthy male and female subjects aged between 18 and 45 years (inclusive) at screening.
* Women of childbearing potential must have a negative serum pregnancy test at screening and a negative urine pregnancy test on Day 1 pre-dose of each treatment period. They must consistently and correctly use a reliable method of contraception, be sexually inactive, or have a vasectomized partner.
* Women of non-childbearing potential (i.e., postmenopausal).
* Body mass index of 18.0 to 32.0 kg/m2 (inclusive) at screening.
* Healthy on the basis of medical history, physical examination, cardiovascular assessments and serology and laboratory tests.
* Previous experience with alcohol consumption and, therefore, familiar with the effects of alcohol.

Exclusion Criteria:

* Pregnant or lactating women.
* Any circumstances or conditions, which, in the opinion of the investigator, may affect full participation in the study or compliance with the protocol.
* Excessive caffeine consumption, defined as ≥ 800 mg per day at screening.
* Nicotine intake within 3 months prior to screening and inability to refrain from nicotine intake from screening until End-of-Study (EOS).
* Previous treatment with any prescribed medications (including vaccines) or over-the-counter (OTC) medications (including herbal medicines such as St John's Wort, homeopathic preparations, vitamins, and minerals) within 2 weeks prior to first study treatment administration.
* History or clinical evidence of alcoholism or drug abuse.
* History of regular alcohol consumption within 6 months of the study defined as an average weekly intake of more than 21 units or an average daily intake of more than 3 units (males), or defined as an average weekly intake of more than 14 units or an average daily intake of more than 2 units (females).
* Individuals of Asian descent or other individuals reporting ethanol intolerance.
* Modified Swiss Narcolepsy Scale total score < 0 at screening or history of narcolepsy or cataplexy.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2018-08-28 (Actual); Primary Completion 2018-10-09 (Actual); Study Completion 2018-10-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline for saccadic peak velocity (degrees/sec) to assess sedation | Several timepoints on Day 1; for up to 24 hours post-dose

OTHER OUTCOMES:
Change from baseline for smooth pursuit (%) to assess eye movement coordination and attention | Several timepoints on Day 1; for up to 24 hours post-dose
Change from baseline for adaptive tracking (%) to assess visuo-motor control and vigilance | Several timepoints on Day 1; for up to 24 hours post-dose
Change from baseline for body sway (antero-posterior in mm / 2 min) to assess postural stability | Several timepoints on Day 1; for up to 24 hours post-dose
Change from baseline for visual analog scales (VAS) Bond & Lader to assess subjective alertness, mood, and calmness | Several timepoints on Day 1; for up to 24 hours post-dose
Change from baseline for VAS for alcohol intoxication to assess subjective effects of ethanol | Several timepoints on Day 1; for up to 24 hours post-dose
ACT-541468 PK endpoints for treatments A and B: Area under the plasma concentration-time curve (AUC) from time zero to 24 h (AUC0-24) | Several timepoints from Day 1 to Day 2 (EOT/EOS); for up to 24 hours post-dose
ACT-541468 PK endpoints for treatments A and B: AUC from zero to infinity (AUC0-∞) | Several timepoints from Day 1 to Day 2 (EOT/EOS); for up to 24 hours post-dose
ACT-541468 PK endpoints for treatments A and B: Maximum plasma concentration (Cmax) | Several timepoints from Day 1 to Day 2 (EOT/EOS); for up to 24 hours post-dose
ACT-541468 PK endpoints for treatments A and B: Time to reach Cmax (tmax) | Several timepoints from Day 1 to Day 2 (EOT/EOS); for up to 24 hours post-dose
ACT-541468 PK endpoints for treatments A and B: Terminal elimination half-life (t½) | Several timepoints from Day 1 to Day 2 (EOT/EOS); for up to 24 hours post-dose
Ethanol PK endpoints for treatments A and C: Breath ethanol concentrations (BrEC) | Several timepoints on Day 1; for up to 24 hours post-dose
Ethanol PK endpoints for treatments A and C: Total ethanol dose (in grams) required to maintain the 0.6 g/L ethanol clamp | Several timepoints on Day 1; for up to 5 hours
Safety endpoints: Treatment-emergent AEs from study treatment administration up to EOT in each treatment period | AEs from Day 1 to Day 2 (EOT/EOS); for up to 2 days post-dose
Safety endpoints: Treatment-emergent SAEs from study treatment administration up to EOT in each treatment period | SAEs from Screening to Safety follow up; for up to 14 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pascale Gasser, Study Director — Idorsia Pharmaceuticals Ltd.
Locations (1):
- Centre For Human Drug Research, Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Berger B, Brooks S, Zuiker R, Richard M, Muehlan C, Dingemanse J. Pharmacological Interactions between the Dual Orexin Receptor Antagonist Daridorexant and Ethanol in a Double-Blind, Randomized, Placebo-Controlled, Double-Dummy, Four-Way Crossover Phase I Study in Healthy Subjects. CNS Drugs. 2020 Dec;34(12):1253-1266. doi: 10.1007/s40263-020-00768-8. Epub 2020 Nov 18. PMID 33205362